CLINICAL TRIAL: NCT04226768
Title: Impact of Enhanced Haematology Palliative Care Services in Patients With Myelodysplastic Syndrome and Acute Myeloid Leukaemia
Brief Title: Enhanced Palliative Care in MDS and AML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Gill Harinder Singh, Harry, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PC001
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic syndrome; Acute myeloid leukemia; Palliative care
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Haematology Palliative Care ("Fast-track") Group (Experimental): Patients who are assigned to enhanced haematology palliative care ("fast-track" group) will be seen, within 2 days of enrollment, at the out-patient clinic or in-patient setting by the haematology palliative care team that comprises a palliative medicine specialist or a haematologist with palliative care experience, a full-time palliative care nurse, and a medical social worker concentrating on haematology palliative patients.
  Interventions: Other: Enhanced Haematology Palliative Care ("Fast-track") Group
- Conventional Supportive Care Group (Active Comparator): Patients who are assigned to the conventional supportive care group will be under care of haematologists and nurse specialists in haematology After 12 weeks of conventional supportive care, patients randomized to this group will receive services from the palliative care team and assessed every two weeks same the "fast-track" group
  Interventions: Other: Conventional Care

INTERVENTIONS:
Other: Enhanced Haematology Palliative Care ("Fast-track") Group — Early and proactive multidisciplinary care
  Arms: Enhanced Haematology Palliative Care ("Fast-track") Group
Other: Conventional Care — Conventional care and referral as indicated
  Arms: Conventional Supportive Care Group

SUMMARY:
Objectives:

The purpose of this study is to evaluate the impact of enhanced haematology palliative care services to the most symptomatic group of blood cancer patients, namely myelodysplastic syndrome (MDS) and acute myeloid leukaemia (AML).

Hypothesis to be tested:

To test whether early integration of dedicated palliative care will improve the quality of life, mood and caregiver burden in patients with MDS and AML.

Design and subjects:

This is a 24-month open-label randomized controlled trial. Subjects include patients with MDS and AML.

Study instruments:

Interventions will be carried out by a dedicated team comprising palliative care physicians, haematologists, palliative care nurse specialists, and social workers. Outcome measures will be determined using validated questionnaires and data collection tools.

Interventions:

In this trial, enhanced haematology palliative care integrated to conventional supportive care versus conventional supportive care alone will be compared.

Main outcome measures:

The primary outcome measures include quality of life, mood and caregiver burden. The secondary outcome measures include number of admissions to acute hospital and intensive care and overall survival.

DETAILED DESCRIPTION:
Acute myeloid leukaemia (AML) and myelodysplastic syndrome (MDS) are heterogeneous haematological malignancies associated with guarded long-term outcomes. In AML, 5-year overall survivals is approximately 40% even in young patients. Relapsed or refractory state is seen in up to 40% of patients with AML is associated with a poor outlook especially in patients in-eligible for intensive treatment. MDS is rarely curable except in young patients eligible for allogeneic haematopoietic stem transplantation (HSCT). MDS failing initial treatment have median survivals of less than 6 months. Most patients with AML and MDS are diagnosed after the age of 65, making them physically-ineligible for intensive curative treatment such as HSCT. In addition to inferior survivals, most patients with relapsed or refractory AML and MDS have profound cytopenia resulting in increased risk of infections and need for frequent blood product support. Quality of life (QOL) is affected due to significant symptom burden, treatment side-effects and repeated admission. Furthermore, an increased caregiver burden could be anticipated. Patients with blood cancers, especially those with AML and MDS experience significant physical and psychological symptoms that are comparable to or exceeding that seen in patients with solid organ cancers.

Well-designed randomized controlled trials have clearly demonstrated the benefits of integrating early palliative care concurrently with standard care in cancer patients. Most of these trials demonstrated improved QOL and mood as well as reduction in the utilization of healthcare services. It is now recommended that in-patients and out-patients with advances malignancies should receive dedicated palliative care services early during the course of the disease. Caregivers may also be referred for palliative services to reduce caregiver burden.

Despite the need for specific palliative care services, growing literature suggests that patients with blood cancer are less likely to receive palliative care services early. We have also shown that most patients with AML receive palliative care late and spend most the end-of-life periods in acute hospitals. In addition, there is a lack of studies examining the impact of early dedicated multidisciplinary palliative care services on blood cancer patients' QOL, mood and caregiver burden.

In this study, investigators designed an open-label randomized controlled-study comparing early enhanced palliative care serviced versus usual care in patients with myelodysplastic syndrome (MDS) and acute myeloid leukaemia (AML).

ELIGIBILITY:
Inclusion Criteria:

1. Myelodysplastic syndrome (MDS) or acute myeloid leukaemia (AML) defined using the World Health Organization Classification 2016.
2. Patients who are able to read and respond to questions in Chinese.

Exclusion Criteria:

Patients who are already receiving care from a palliative care unit will be excluded. Patients who require immediate palliative care service, e.g. end-of-life care, will be excluded and receive palliative care immediately.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
McGill Quality of Life (MQOL) Questionnaire Score | 24 weeks
  It is a 17-item patient-rated measure of QOL for patients receiving palliative care.This questionnaire was translated and validated in Hong Kong. The questionnaire consists of five domains: physical well-being (five items), psychological well-being (six items), existential well-being (four items), support (two items), and sexual function (one item). In addition, there is a single item to rate their perceived quality of life. The response categories are based on a numerical scale from 0-10 with verbal anchors at the end of the scale. For the final statistical analysis, all scores are transposed on a 0-10 scale, with 0 representing the least and 10 indicating the most desirable situation. The mean total QOL score is the average of all the 5 domain scores, with 0 representing the worst situation. The overall validation results of the MQOL-HK were acceptable. Cronbach's α for the MQOL-HK subscale ranged from 0.68 to 0.85.
Hospital Anxiety and Depression Scale (HADS) | 24 weeks
  Levels of anxiety and depression were self-rated by HADS, which has been found to perform well as a test for such symptoms in the general population, in cancer patients and in primary care patients. Subjects decide on how each item applies to them on a scale ranging from no feelings of anxiety or depression (0) to severe feelings of anxiety or depression (3), with scores ranging from 0 to 21 on each subscale. A subscale score of 8 to 10 indicates a possible case of anxiety or depression, whereas a subscale score of 11 or higher indicates a definite case of anxiety or depression. Severe depression or anxiety disorders are suspected for subjects scoring 15 or higher.24 The Cantonese-Chinese version of the HADS25 has been found to have good internal consistency (Cronbach's α=0.77), reasonable sensitivity (0.79) and specificity (0.80), as well as positive (0.77) and negative predictive values (0.82).
Zariet Burden Interview (ZBI) | 24 weeks
  The ZBI is a widely used 22-item assessment tool for measuring the caregiver's perceived burden in providing family care. The questionnaire was translated, and modified according to Hong Kong cultural standards.
  The ZBI scale was developed to measure burden among family caregivers of persons with dementia; however, it has been used in other populations and was selected for this study because of the high reliability and validity of the Chinese version, indicated by a Cronbach's alpha of 0.99 and a correlation coefficient of 0.81. The correlation between ZBI and general Health Questionnaire was 0.59 (p<0.001), and the correlation between Caregiver Activity Survey was 0.057 (p<0.001), suggesting high conceptual validity.
  The items were scored on a five-point scale ranging from 0 (never) to 4 (always). Scores were calculated by summing up the total chosen statement which ranges from 0 to 88, that higher scores implying greater perceived caregiver burden.

SECONDARY OUTCOMES:
Number of admissions to acute hospital | 24 weeks
  Number
Number of admission to intensive care unit | 24 weeks
  Number
Overall survival | 24 weeks
  Time (in weeks) from the data of recruitment to death or latest follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Singh Harry Gill, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, the University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Result] Thol F, Schlenk RF, Heuser M, Ganser A. How I treat refractory and early relapsed acute myeloid leukemia. Blood. 2015 Jul 16;126(3):319-27. doi: 10.1182/blood-2014-10-551911. Epub 2015 Apr 7. PMID 25852056
- [Result] Juliusson G, Antunovic P, Derolf A, Lehmann S, Mollgard L, Stockelberg D, Tidefelt U, Wahlin A, Hoglund M. Age and acute myeloid leukemia: real world data on decision to treat and outcomes from the Swedish Acute Leukemia Registry. Blood. 2009 Apr 30;113(18):4179-87. doi: 10.1182/blood-2008-07-172007. Epub 2008 Nov 13. PMID 19008455
- [Result] Prebet T, Gore SD, Esterni B, Gardin C, Itzykson R, Thepot S, Dreyfus F, Rauzy OB, Recher C, Ades L, Quesnel B, Beach CL, Fenaux P, Vey N. Outcome of high-risk myelodysplastic syndrome after azacitidine treatment failure. J Clin Oncol. 2011 Aug 20;29(24):3322-7. doi: 10.1200/JCO.2011.35.8135. Epub 2011 Jul 25. PMID 21788559
- [Result] Epstein AS, Goldberg GR, Meier DE. Palliative care and hematologic oncology: the promise of collaboration. Blood Rev. 2012 Nov;26(6):233-9. doi: 10.1016/j.blre.2012.07.001. Epub 2012 Aug 5. PMID 22874874
- [Result] Manitta V, Zordan R, Cole-Sinclair M, Nandurkar H, Philip J. The symptom burden of patients with hematological malignancy: a cross-sectional observational study. J Pain Symptom Manage. 2011 Sep;42(3):432-42. doi: 10.1016/j.jpainsymman.2010.12.008. Epub 2011 Apr 7. PMID 21477979
- [Result] Fadul NA, El Osta B, Dalal S, Poulter VA, Bruera E. Comparison of symptom burden among patients referred to palliative care with hematologic malignancies versus those with solid tumors. J Palliat Med. 2008 Apr;11(3):422-7. doi: 10.1089/jpm.2007.0184. PMID 18363482
- [Result] Manitta VJ, Philip JA, Cole-Sinclair MF. Palliative care and the hemato-oncological patient: can we live together? A review of the literature. J Palliat Med. 2010 Aug;13(8):1021-5. doi: 10.1089/jpm.2009.0267. PMID 20712465
- [Result] Ferrell BR, Temel JS, Temin S, Alesi ER, Balboni TA, Basch EM, Firn JI, Paice JA, Peppercorn JM, Phillips T, Stovall EL, Zimmermann C, Smith TJ. Integration of Palliative Care Into Standard Oncology Care: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2017 Jan;35(1):96-112. doi: 10.1200/JCO.2016.70.1474. Epub 2016 Oct 28. PMID 28034065
- [Result] Bakitas M, Lyons KD, Hegel MT, Balan S, Brokaw FC, Seville J, Hull JG, Li Z, Tosteson TD, Byock IR, Ahles TA. Effects of a palliative care intervention on clinical outcomes in patients with advanced cancer: the Project ENABLE II randomized controlled trial. JAMA. 2009 Aug 19;302(7):741-9. doi: 10.1001/jama.2009.1198. PMID 19690306
- [Result] Bakitas MA, Tosteson TD, Li Z, Lyons KD, Hull JG, Li Z, Dionne-Odom JN, Frost J, Dragnev KH, Hegel MT, Azuero A, Ahles TA. Early Versus Delayed Initiation of Concurrent Palliative Oncology Care: Patient Outcomes in the ENABLE III Randomized Controlled Trial. J Clin Oncol. 2015 May 1;33(13):1438-45. doi: 10.1200/JCO.2014.58.6362. Epub 2015 Mar 23. PMID 25800768
- [Result] Dionne-Odom JN, Azuero A, Lyons KD, Hull JG, Tosteson T, Li Z, Li Z, Frost J, Dragnev KH, Akyar I, Hegel MT, Bakitas MA. Benefits of Early Versus Delayed Palliative Care to Informal Family Caregivers of Patients With Advanced Cancer: Outcomes From the ENABLE III Randomized Controlled Trial. J Clin Oncol. 2015 May 1;33(13):1446-52. doi: 10.1200/JCO.2014.58.7824. Epub 2015 Mar 23. PMID 25800762
- [Result] Zimmermann C, Swami N, Krzyzanowska M, Hannon B, Leighl N, Oza A, Moore M, Rydall A, Rodin G, Tannock I, Donner A, Lo C. Early palliative care for patients with advanced cancer: a cluster-randomised controlled trial. Lancet. 2014 May 17;383(9930):1721-30. doi: 10.1016/S0140-6736(13)62416-2. Epub 2014 Feb 19. PMID 24559581
- [Result] LeBlanc TW, El-Jawahri A. When and why should patients with hematologic malignancies see a palliative care specialist? Hematology Am Soc Hematol Educ Program. 2015;2015:471-8. doi: 10.1182/asheducation-2015.1.471. PMID 26637760
- [Result] Cheng HW, Li CW, Chan KY, Au HY, Chan PF, Sin YC, Szeto Y, Sham MK. End-of-life characteristics and palliative care provision for elderly patients suffering from acute myeloid leukemia. Support Care Cancer. 2015 Jan;23(1):111-6. doi: 10.1007/s00520-014-2333-x. Epub 2014 Jul 5. PMID 24996833
- [Result] Cheng HW. Optimizing End-of-Life Care for Patients With Hematological Malignancy: Rethinking the Role of Palliative Care Collaboration. J Pain Symptom Manage. 2015 May;49(5):e5-6. doi: 10.1016/j.jpainsymman.2015.01.008. Epub 2015 Feb 2. No abstract available. PMID 25656326
- [Result] Roberts C, Torgerson D. Randomisation methods in controlled trials. BMJ. 1998 Nov 7;317(7168):1301. doi: 10.1136/bmj.317.7168.1301. No abstract available. PMID 9804722
- [Result] Rinck GC, van den Bos GA, Kleijnen J, de Haes HJ, Schade E, Veenhof CH. Methodologic issues in effectiveness research on palliative cancer care: a systematic review. J Clin Oncol. 1997 Apr;15(4):1697-707. doi: 10.1200/JCO.1997.15.4.1697. PMID 9193371
- [Result] Higginson IJ, Finlay IG, Goodwin DM, Hood K, Edwards AG, Cook A, Douglas HR, Normand CE. Is there evidence that palliative care teams alter end-of-life experiences of patients and their caregivers? J Pain Symptom Manage. 2003 Feb;25(2):150-68. doi: 10.1016/s0885-3924(02)00599-7. PMID 12590031
- [Result] Chan KY, Yip T, Yap DY, Sham MK, Wong YC, Lau VW, Li CW, Cheng BH, Lo WK, Chan TM. Enhanced Psychosocial Support for Caregiver Burden for Patients With Chronic Kidney Failure Choosing Not to Be Treated by Dialysis or Transplantation: A Pilot Randomized Controlled Trial. Am J Kidney Dis. 2016 Apr;67(4):585-92. doi: 10.1053/j.ajkd.2015.09.021. Epub 2015 Nov 6. PMID 26549852
- [Result] Lo RS, Woo J, Zhoc KC, Li CY, Yeo W, Johnson P, Mak Y, Lee J. Cross-cultural validation of the McGill Quality of Life questionnaire in Hong Kong Chinese. Palliat Med. 2001 Sep;15(5):387-97. doi: 10.1191/026921601680419438. PMID 11591090
- [Result] Leung CM, Wing YK, Kwong PK, Lo A, Shum K. Validation of the Chinese-Cantonese version of the hospital anxiety and depression scale and comparison with the Hamilton Rating Scale of Depression. Acta Psychiatr Scand. 1999 Dec;100(6):456-61. doi: 10.1111/j.1600-0447.1999.tb10897.x. PMID 10626925
- [Result] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Result] Arai Y, Kudo K, Hosokawa T, Washio M, Miura H, Hisamichi S. Reliability and validity of the Japanese version of the Zarit Caregiver Burden interview. Psychiatry Clin Neurosci. 1997 Oct;51(5):281-7. doi: 10.1111/j.1440-1819.1997.tb03199.x. PMID 9413874
- [Result] Ko KT, Yip PK, Liu SI, Huang CR. Chinese version of the Zarit caregiver Burden Interview: a validation study. Am J Geriatr Psychiatry. 2008 Jun;16(6):513-8. doi: 10.1097/JGP.0b013e318167ae5b. PMID 18515696
- [Result] Kimmel PL, Emont SL, Newmann JM, Danko H, Moss AH. ESRD patient quality of life: symptoms, spiritual beliefs, psychosocial factors, and ethnicity. Am J Kidney Dis. 2003 Oct;42(4):713-21. doi: 10.1016/s0272-6386(03)00907-7. PMID 14520621